CLINICAL TRIAL: NCT04668508
Title: A Phase II Study of Anlotinib Combined With Radiation in Patients With Malignant Brainstem Glioma
Brief Title: Anlotinib to Malignant Brainstem Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-217
Record Dates: First submitted 2020-11-26; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Malignant Brain Stem Tumor; Glioma
MeSH Terms: conditions — Glioma | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: Anlotinib combined with radiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib combined with radiation (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — concurrent using anlotinib combined with radiation plus adjuvant anlotinib after radiotherapy until disease progress or develop into serious adverse events.

SUMMARY:
This study is a single-arm, open-label, phase II study of anlotinib combined with radiation in the treatment of patients with malignant brainstem glioma. Twenty five patients will be enrolled in the study who is diagonsis with malignant brainstem glioma. The primary objective includes disease control rate (DCR), the role of antinib combined with radiotherapy in improving quality of life and 6-month progression-free survival rate. The secondary objective include overall survival (OS), toxicity profile. Exploratory objectives include the use of plasma specimens and cerebrospinal fluid (if possible) to detect biomarkers predicting the efficacy of anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before any trial-related processes are implemented;
2. Age ≥ 18 years old and ≤ 70 years old;
3. Life expectancy exceeds 3 months;
4. The investigator confirmed at least one measurable lesion according to the RECIST 1.1 standard. A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if it is confirmed to have progressed;
5. Patients with WHO Ⅲ - Ⅳ brain stem glioma confirmed by histology or radiology;
6. The Karnofsky score has to >40;
7. For subjects who had undergone surgical biopsy or treatment, the surgical incision has to be healed well;
8. No prior radiotherapy, chemotherapy, immunotherapy or biotherapy has been performed;
9. Hematological function is sufficient, defined as absolute neutrophil count

   ≥1.5×109 /L, platelet count ≥100 ×109 /L, hemoglobin ≥90g/L (no history of blood transfusion within 7 days);
10. Hepatic function is adequate, defined as all patients with total bilirubin levels ≤ 1.5 times normal upper limit (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN, or for patients with liver metastases , AST and ALT levels ≤ 5 times ULN;
11. adequate renal function, defined as creatinine clearance ≥ 45 ml / min (Cockcroft-Gault formula);
12. Coagulation function is adequate, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulant therapy, as long as the INR or PT is within the range of anticoagulant drugs can;
13. Female subjects of childbearing age should be negative for urine or serum pregnancy test within 3 days prior to receiving the first study drug. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required;
14. If there is a risk of conception, male and female patients need to use high-efficiency contraception (ie, an annual failure rate of less than 1%) and continue until at least 180 days after stopping the trial treatment; Note: If abstinence is normal for the subject Lifestyle and preferred methods of contraception can be used as a method of contraception.

Exclusion Criteria:

1. WHO grade I-II glioma or imaging diagnosis of low-level brainstem glioma;
2. Supratentorial gliomas in adults involve the brain stem;
3. Patients with contraindications for MRI;
4. Patients with any signs or history of bleeding physique;
5. Currently participating in interventional clinical research treatment, or receiving other research drugs or research equipment within 4 weeks prior to the first dose;
6. Severe intracranial infection;
7. Any arterial thrombosis, embolism or ischemia occurred within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within 3 months prior to enrollment (implanted IV port or catheter-derived thrombosis, or superficial vein thrombosis is not considered a "serious" thrombosis embolism);
8. Prior or concurrent malignancies excepting for adequately treated skin cancer (non-melanoma), in situ cervical carcinoma or cured malignant disease≥5 years;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
disease control rate | through study completion, an average of 1 year
  based on RECIST1.1
6-month progression-free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, assessed up to 6 months
  proportion of patients with progression-free survival longer than 6 months.
6-month quality of life deterioration-free survival | From date of randomization until the date of first documented progression or date of death from any cause, assessed up to 6 months
  quality of life

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of first documented progression or date of death from any cause, assessed up to 6 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided